CLINICAL TRIAL: NCT04915859
Title: Semiconductor Heat Extraction Cooling During and After Exercise in the Heat
Brief Title: Semiconductor Heat Extraction Cooling
Acronym: SHE-Cool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Kelvi - Hypothermia Devices, Inc. (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H21-0031
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants will receive four cooling treatment on separate study visits 1)hand cooling at 12-15C 2)hand cooling at 16-20C 3)passive cooling 4)back and hand cooling (at 12-15C or 16-20C depending on results of trials 1-3)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cooling (Active Comparator): Participants will be actively cooled during rest breaks
  Interventions: Other: Hand Cooling at 12-15 degrees celsius; Other: Hand Cooling at 16-20 degrees celsius; Other: hand and back cooling at 12-15 or 16-20 degrees celsius
- No Intervention (Placebo Comparator): Participants will participate in "passive cooling" where they sit in a chair during rest
  Interventions: Other: Passive cooling

INTERVENTIONS:
Other: Hand Cooling at 12-15 degrees celsius — hand cooling at 12-15 degrees celsius will be performed for active cooling by having participants place their hands on the cooling device set to this temperature
  Arms: Active Cooling
Other: Hand Cooling at 16-20 degrees celsius — hand cooling at 16-20 degrees celsius will be performed for active cooling by having participants place their hands on the cooling device set to this temperature
  Arms: Active Cooling
Other: hand and back cooling at 12-15 or 16-20 degrees celsius — hand and back cooling at 12-15 or 16-20 degrees celsius will be performed for active cooling by having participants place their hands on the cooling device set to this temperature while also wearing the back wrap cooling device set to this temperature
  Arms: Active Cooling
Other: Passive cooling — participants will sit in a chair and "passively cool" (no active intervention)
  Arms: No Intervention

SUMMARY:
Heat-related injuries and other physiological stresses continue to be a significant threat to the health and operational effectiveness of the US Armed Forces (Armed Forces Health Surveillance 2011). This is because military personnel are exposed to exertional and environmental heat-stress factors during both deployment and training at US installations in hot and humid climates. Cold water immersion (CWI) is considered the gold standard for the treatment of exertional heat stroke (EHS) and has been shown to increase survival rates to 100% with the implementation of CWI best practices. However, in a field setting other cooling strategies have been developed to aid in the prevention of EHS and other heat-related illnesses. One such proposed strategy is a portable hand cooling device that does not require the use of ice or water. Therefore, the primary purpose of this investigation is to validate hand and back cooling devices using physiological, cognitive, performance, and perceptual responses that occur during and following rest, exercise, and cooling in the heat.

ELIGIBILITY:
Inclusion Criteria:

* male or female between the ages of 18-45 years
* females only: taking monophasic birth control pill this is to maintain applicability to a large portion of the female population that take birth control and limit the influence of varying estrogen and progesterone levels throughout the menstrual cycle. during the informational session researchers will have this list of brands of monophasic birth control pill brands to determine if the participant is eligible Brevicon Modicon Wera Balziva Gildagia Philith Zenchent Estarylla Previfem Sprintec Ocella Yasmin Zarah Yaz Safyral Beyaz Cryselle Elinest Ogestrel Apri Desogen Juleber Reclipsen Solia Levora Altavera Daysee Lessina Lybrel Amethia Jolessa all trials will only be conducted during the days the participant is on the hormone pill (not on the days during which they are taking the placebo pill)
* been cleared by the medical monitor for this study
* VO2max > 45ml/kg/min (measure obtained only from the VO2max test performed on the treadmill on Visit 1)
* Aerobically active (at least 30 minutes of aerobic exercise 4-5 days per week)

Exclusion Criteria:

* Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
* Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
* Fever or current illness at the time of testing
* History of cardiovascular, metabolic, or respiratory disease
* A family member died for no apparent reason, had a heart attack, died from heart problems, or sudden death before the age of 50
* Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin)
* Have a history of heat related illness
* Have any allergies or adverse reactions to the cold (e.g. Cold Uticaria, Raynauds -Phenomenon/Disease, or Cryoglobulinanemia)
* Have claustrophobia or feelings of discomfort towards sitting in a small, enclosed area
* Have allergies to medical and/or adhesive tape
* Have eating disorders
* History of COVID-19 unless cleared by a physician for exercise at the level exercise required to participate in this study. The physician must be made aware of what is required to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in VO2max between Cycle ergometer and treadmill | through study completion, an average of 2 weeks
  Participants will be fitted with a Hans Rudolph mask attached to a breathing tube to measure the expired air delivered to the metabolic cart system during the exercise protocol. The metabolic cart will continuously measure oxygen consumption (VO2) to asess their VO2max value.
Metabolic Heat Production | through study completion, an average of 2 weeks
  Participants will be tested for 3-5 minutes at different % of their VO2max. It will include 5 stages.
Change in Rectal Temperature | through study completion, an average of 2 weeks
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Heart Rate | through study completion, an average of 2 weeks
  A heart rate monitor will be worn by participant throughout exercise/cooling protocol
Change in Mean Skin temperature | through study completion, an average of 2 weeks
  Prior to the start of exercise, participants will be instrumented with iButton skin temperature sensors on the chest, arm, thigh, calf, back of hand, and ankle
Change in Rating of Perceived Exertion | through study completion, an average of 2 weeks
  6-20 scale that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.
Change in Performance Measures | through study completion, an average of 2 weeks
  Participants will perform a performance battery consisting of a wingate anaerobic power test, grip strength test, and broad jump test
Change Injury Risk Assessment Measures | through study completion, an average of 2 weeks
  Participants will perform a injury risk assessment battery consisting of a balance and squat form assessments
Change in Cognitive Measures | through study completion, an average of 2 weeks
  Participants will perform 2 cognitive tests (Go-Nogo and Stroop) on a laptop to measure reaction time and errors. Both tests should take 5 minutes
Change in Recovery | through study completion, an average of 2 weeks
  Participants will be provided a WHOOP strap and Polar heart rate strap at their first visit. They will be instructed on how to download the associated apps and how to charge and care for the devices. They will be provided instructions with how to take heart rate measures. The WHOOP and heart rate measures will provide data on sleep quality and quantity, strain, and recovery.

SECONDARY OUTCOMES:
Change in Thermal Sensation | through study completion, an average of 2 weeks
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot
Change in Perception of Fatigue | through study completion, an average of 2 weeks
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).
Change in Perception of thirst | through study completion, an average of 2 weeks
  0-9 (no thirst to extreme thirst) Scale that indicates how thirsty the subject feels. A higher score is considered a negative outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Korey Stringer Institute, University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No